CLINICAL TRIAL: NCT07343115
Title: Familial Systemic Scleroderma
Acronym: SCLERO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9820
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Systemic Scleroderma
Keywords: Systemic Scleroderma; Familial Systemic Scleroderma; Autoimmune disease
MeSH Terms: conditions — Scleroderma, Systemic; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Studying familial forms of systemic scleroderma offers several advantages:

1. To better understand the pathophysiology of a complex autoimmune disease based on "extreme" cases (familial forms);
2. To identify potential molecular markers predictive of disease progression;
3. To identify potential pathophysiological targets for developing new therapies, particularly relevant in severe and refractory forms of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (≥ 18 years of age)
* Subjects diagnosed with systemic scleroderma by a clinician (including limited, diffuse, and sine scleroderma SSc, as well as overlap syndromes with myositis) and meeting at least the VEDOSS criteria: Raynaud's phenomenon + 1 other criterion from among: sausage fingers, antinuclear antibodies, scleroderma-specific antibodies (anti-centromere, anti-RNApolIII, anti-ScL70), capillaroscopic abnormalities
* At least one first-degree relative with systemic scleroderma meeting the same criteria

Exclusion Criteria:

- Subject who has expressed opposition to participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects diagnosed with systemic scleroderma by a clinician
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
Description of the clinical characteristics of patients with familial systemic scleroderma | Up to 12 months
  The clinical presentation describes how the disease manifests in patients:
  the symptoms, their severity, and their progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine interne et Immunologie clinique - CHU de Strasbourg - France, Strasbourg, France